CLINICAL TRIAL: NCT01047865
Title: Recurrence of T1D in Pancreas Transplantation
Brief Title: Type 1 Diabetes Recurrence in Pancreas Transplants
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, George W. Burke, Professor of Surgery, University of Miami
Other Study IDs: 20053039
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes (T1D); Autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreas-kidney transplant: pancreas-kidney transplant recipients with type 1 diabetes.

SUMMARY:
The hypothesis is that humoral and cellular islet-specific responses are an early risk factor for recurrence of autoimmunity and hyperglycemia in simultaneous pancreas-kidney (SPK) recipients independent of alloimmunity. This study will test the hypothesis and will assess their individual and combined predictive value.

DETAILED DESCRIPTION:
To identify the factors associated with recurrence of diabetes in subjects who received a simultaneous pancreas-kidney (SPK) or pancreas transplant. The study will see if there are changes in the participant's blood that will help the investigator know whether diabetes has returned after the transplant.

SPK patients will be retrospectively analyzed to determine frequency, levels and time course of autoantibody recurrence and predictive value of autoantibodies for recurrence of the disease.

This study will prospectively follow our existing and our new pancreas transplant recipients to monitor autoantibody levels, monitor and phenotype autoreactive T cells in peripheral blood. This will happen monthly for 24 months.

This study will assess the presence or absence of insulitis in the transplanted pancreas from biopsies performed in recipients with consistent recurrence of multiple autoantibodies.

It will also monitor and phenotype autoreactive T cells from the pancreatic infiltrate obtained by pancreatic transplant biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed and has signed a dated IRB approval informed consent form and is willing to follow study procedures for the extent of the study (24 months). Parent or legal guardian must provide written consent for patients <18 years of age.
* Age 18-75 years.
* Recipient of simultaneous pancreas and kidney transplant
* Primary or secondary renal allograft: living or deceased

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a pancreas-kidney.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes who received a simultaneous pancreas-kidney (SPK) transplant
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2005-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Retrospective and prospective analysis of pancreas transplant recipients to determine frequency, and time course of autoantibody recurrence of disease. Prospective follow up to: monitor autoantibody levels, monitor and phenotype autoreactive T | up to 5 years
  Antibody recurrence

SECONDARY OUTCOMES:
Monitor autoantibody levels as well as phenotype autoreactive T cells in peripheral blood. | up to 15 years
  Antibodies levels

CONTACTS AND LOCATIONS:
Overall Officials: George Burke, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine Transplant Clinic, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vendrame F, Hopfner YY, Diamantopoulos S, Virdi SK, Allende G, Snowhite IV, Reijonen HK, Chen L, Ruiz P, Ciancio G, Hutton JC, Messinger S, Burke GW 3rd, Pugliese A. Risk Factors for Type 1 Diabetes Recurrence in Immunosuppressed Recipients of Simultaneous Pancreas-Kidney Transplants. Am J Transplant. 2016 Jan;16(1):235-45. doi: 10.1111/ajt.13426. Epub 2015 Aug 28. PMID 26317167
- [Result] Burke GW 3rd, Vendrame F, Virdi SK, Ciancio G, Chen L, Ruiz P, Messinger S, Reijonen HK, Pugliese A. Lessons From Pancreas Transplantation in Type 1 Diabetes: Recurrence of Islet Autoimmunity. Curr Diab Rep. 2015 Dec;15(12):121. doi: 10.1007/s11892-015-0691-5. PMID 26547222
- [Result] Pugliese A, Vendrame F, Reijonen H, Atkinson MA, Campbell-Thompson M, Burke GW. New insight on human type 1 diabetes biology: nPOD and nPOD-transplantation. Curr Diab Rep. 2014 Oct;14(10):530. doi: 10.1007/s11892-014-0530-0. PMID 25142715
- [Result] Pugliese A, Yang M, Kusmarteva I, Heiple T, Vendrame F, Wasserfall C, Rowe P, Moraski JM, Ball S, Jebson L, Schatz DA, Gianani R, Burke GW, Nierras C, Staeva T, Kaddis JS, Campbell-Thompson M, Atkinson MA. The Juvenile Diabetes Research Foundation Network for Pancreatic Organ Donors with Diabetes (nPOD) Program: goals, operational model and emerging findings. Pediatr Diabetes. 2014 Feb;15(1):1-9. doi: 10.1111/pedi.12097. Epub 2013 Dec 10. PMID 24325575
- [Result] Ciancio G, Sageshima J, Chen L, Gaynor JJ, Hanson L, Tueros L, Montenora-Velarde E, Gomez C, Kupin W, Guerra G, Mattiazzi A, Fornoni A, Pugliese A, Roth D, Wolf M, Burke GW 3rd. Advantage of rapamycin over mycophenolate mofetil when used with tacrolimus for simultaneous pancreas kidney transplants: randomized, single-center trial at 10 years. Am J Transplant. 2012 Dec;12(12):3363-76. doi: 10.1111/j.1600-6143.2012.04235.x. Epub 2012 Sep 4. PMID 22946986